CLINICAL TRIAL: NCT03070431
Title: High-precision Radiotherapy of Motor Deficits Due to Metastatic Spinal Cord Compression
Acronym: PRE-MODE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Prof. Dirk Rades, MD, Professor Dr. med., University Hospital Schleswig-Holstein
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRE-MODE
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Results first posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Spinal Cord Compression Due to Metastasis to Spine
Keywords: spinal cord compression, radiotherapy
MeSH Terms: conditions — Spinal Cord Compression

STUDY DESIGN:
Intervention Model Description: Single arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-precision RT 5x5 Gy in 1 week (Experimental): Patients with motor deficits of the lower extremities due to metastatic spinal cord compression (MSCC) will receive 5x5 Gy of high-precision RT in 1 week.
  Interventions: Radiation: High-precision RT 5x5 Gy in 1 week

INTERVENTIONS:
Radiation: High-precision RT 5x5 Gy in 1 week — Patients included in this study will receive a high-precision radiotherapy with 5x5 Gy in 1 week

SUMMARY:
The major goal of this clinical study is to investigate to which extent high-precision radiotherapy (RT) with modern techniques can prevent progression or recurrence of motor deficits (weakness) of the legs following RT. In addition, it will be evaluated to which extent RT can lead to improvement of motor function, ambulatory status, sensory function and sphincter dysfunction, to pain relief and to improvement in quality of life, side effects and overall survival. For this purpose 44 patients who will receive modern high-precision RT treatment for the metastases on their vertebral bodies will be included into this phase 2 study. The results of the high-precision RT with a treatment of 5x5 Gray (Gy) in 1 week will be compared to data of a historical control group. The data set of the historical control group consists of more than 500 patients who received conventional RT with 5x4 Gy. The data collected in 1 week treatment will be compared. It is intended to show superiority regarding the local progression-free survival (LPFS) for the high-precision RT when compared with the conventional RT.

DETAILED DESCRIPTION:
This is a multinational, multicenter study (single arm) supplemented by a comparison to a historical, propensity score matched control group (superiority study).

A total of 44 patients (40 patients + 10% for potential drop-outs) who will receive modern high-precision radiotherapy (RT) treatment for the metastases on their vertebral bodies are planned to take part in the clinical study. The historical control group treated with 5x4 Gy of conventional RT between 2001 and 2016 consists of more than 500 patients The primary aim of this study is to investigate the local progression-free survival (LPFS) of metastatic spinal cord compression (MSCC) after 5x5 Gray (Gy) of high-precision RT and to demonstrate that this regimen results in significantly better 6-month LPFS than conventional RT with 5x4 Gy. For the high-precision RT volumetric modulated arc therapy (VMAT), stereotactic body radiotherapy (SBRT) is allowed for treatment of patients with involvement of only one vertebra, if the required constraints can be met. LPFS is defined as freedom from progression of motor deficits during RT and freedom from an in-field recurrence of MSCC (i.e. freedom from motor deficits due to a recurrence of MSCC in the previously irradiated parts of the spine) following RT. The LPFS rate will be assessed 6 months after the end of RT.

In patients treated with RT alone for MSCC, conventional RT with 10x3 Gy in 2 weeks results in similar motor function but significantly better LPFS than conventional RT with 5x4 Gy in 1 week. Since patients with MSCC are often significantly impaired, a RT regimen with an overall treatment time of only 1 week would be preferable if it resulted in similar LPFS as 10x3 Gy in 2 weeks. This may be achieved with 5x5 Gy in 1 week, since the equivalent dose in 2 Gy fractions (EQD2) with respect to tumor cell kill of 5x5 Gy and 10x3 Gy are similar. The tolerance dose of the spinal cord, 5x5 Gy can be safely administered with high-precision RT such as VMAT (or SBRT). Therefore, the present study investigates the LPFS after high-precision RT with 5x5 Gy in 1 week. To demonstrate superiority the patients of this study will be compared to a historical control group receiving conventional RT with 5x4 Gy in 1 week. If superiority regarding LPFS can be shown for high-precision RT with 5x5 Gy, patients with MSCC would benefit from this regimen, since they can achieve high LPFS rates with an RT regimen lasting only 1 week (5x5 Gy) instead of 2 weeks (10x3 Gy). This study aims to make a significant contribution to the most appropriate RT schedule for patients with MSCC.

In accordance with a previous study assessing local control of MSCC, the following patient characteristics will be recorded to allow adequate comparison with the historical, propensity-score matched control group:

* Age (2 groups, depending on median age)
* Gender
* Type of primary tumor (breast cancer vs. prostate cancer vs. myeloma/lymphoma vs. lung cancer vs. other tumors)
* Interval from tumor diagnosis to MSCC (≤15 months vs. >15 months)
* Number of involved vertebrae (1-2 vs. ≥3)
* Other bone metastases at the time of RT (no vs. yes)
* Visceral metastases at the time of RT (no vs. yes)
* Time developing motor deficits prior to RT (1-7 days vs. 8-14 days vs. >14 days)
* Ambulatory status prior to RT (no vs. yes)
* Eastern Cooperative Oncology Group (ECOG) performance score (1-2 vs. 3-4) Study arm: 5x5 Gy of high-precision RT in 1 week Historical control: 5x4 Gy of conventional RT in 1 week Follow-up directly and at 1, 3 and 6 months following RT RT is administered as high-precision RT with 25.0 Gy in 1 week, i.e. with 5.0 Gy per fraction on 5 days per week (representing an EQD2 of 43.8 Gy for radiation myelopathy). An EQD2 of 45 Gy is estimated to be associated with a risk of radiation-related myelopathy of 0.03% and is therefore considered safe. The clinical target volume (CTV) includes the vertebral and soft tissue tumor as seen on the planning computed tomography and diagnostic MR-imaging, the spinal canal, the width of the involved vertebrae, and half a vertebra above and below those vertebrae involved by MSCC. The planning target volume (PTV) should include the CTV plus 0.8 cm and should be covered by the 95%-isodose. The maximum relative dose allowed to the spinal cord is 101.5% of the prescribed dose (representing an EQD2 of 44.9 Gy for radiation myelopathy). This maximum dose is estimated to be associated with a risk of radiation-related of <0.03% and is, therefore, also considered safe. Both the EQD2 of the prescribed dose (41.7 Gy) and the EQD2 of the maximum dose (43.8 Gy) are well below the tolerance dose of bone. In accordance with the Quantitative Analyses of Normal Tissue Effects in the Clinic (QUANTEC) data, the mean doses EQD2 for esophagus, heart and lung must be <34 Gy, <26 Gy and ≤7 Gy, respectively. Taking into account a radiation regimen of five fractions, the corresponding mean doses per fraction are 4.5 Gy, 3.8 Gy and 1.54 Gy, respectively. MSCC may affect single or multiple spinal sites. All sites need to be treated with high-precision RT following the dose prescriptions and constraints given above.

It is recommended that the patients receive concomitant treatment with dexamethasone during the period of radiotherapy if indicated.

Quality assurance plan:

Monitoring: The Centre for Clinical Trials Lübeck will conduct clinical on-site monitoring at the German sites according to Good Clinical Practice and written standard operating procedures (SOPs) to ensure the patients' rights and safety as well as the reliability of trial results.

The frequency of monitoring visits per site will be defined depending on the recruitment rate and the quality of data.

Patient Registration:

The patients were assigned 2 code numbers, the number of the contributing center plus a patient identification number starting with 001 and chronologically ongoing.

Coordination and supervision of the inclusion of the patients will be performed by the Department of Radiation Oncology of the University of Lübeck, Germany.

Sample size calculation:

The primary goal of this study is to assess high-precision RT with 5x5 Gy in 1 week with respect to 6-month LPFS and to demonstrate that this rate is superior to conventional RT with 5x4 Gy with respect to LPFS of MSCC (hypothesis).

With respect to tumor cell kill, the EQD2 of 5x5 Gy is similar to the EQD2 of 10x3 Gy (31.3 Gy vs. 32.5 Gy) and higher than the EQD2 of 5x4 Gy (23.3 Gy) . In a previous prospective non-randomized study, the 6-month LPFS rates were 86% after longer-course RT and 67% after short-course RT, respectively (p=0.034). In that study, 95 of 117 patients (81%) in the longer-course RT group had received 10x3 Gy, and 91 of 114 patients (80%) in the short-course RT group had received 5x4 Gy. Thus, assuming - for the present study - that conventional RT with 5x4 Gy in fact results in a 6-month LPFS rate of 67%, an increase by roughly 20 percentage point is considered to be clinically minimal relevant and even appears to be realistic when applying high-precision RT with 5x5 Gy.

The sample size is chosen to obtain prospective data that can be interpreted on its own and to allow for comparison with historical data:

* A sample size of at least 40 eligible patients is needed to estimate the probability of LPFS at 6 month with adequate precision, based on the following assumptions:

  * 6-month LPFS can be assumed to be 87%
  * 6-month LPFS is to be estimated with a precision of plus/minus 20 percentage points expressed as the half length of the associated two-sided confidence interval with a confidence coefficient of 95%.
  * The power -i.e. the probability to obtain this precision, should be at least 80%
  * Confidence limits are used as the approach for sample size. Assuming that roughly 10% of enrolled patients will not be eligible for efficacy analysis due to early lost-to-follow-up or due to premature discontinuation of high-precision RT, a total of 44 patients should be enrolled in the prospective part of the trial.
* The aim of the confirmatory study is to compare the prospectively collected data with a historical, propensity-score matched cohort collected up to the time of data analysis. Assuming for simplicity and conservative power calculation that this comparison could be conducted with a simple Pearson-Chi-Square test using a two-sided significance level of 5% (10%), a power of 79% (86%) is reached, if 40 patients are treated with high-precision RT and roughly 400 patients of the historical control group qualify for Propensity-Score adjusted comparison and assuming that the expected 6-month LPFS are 87% and 67%, respectively. Taking into account that the more sophisticated propensity-score adjusted statistical analysis will increase statistical power, the power for treatment arm comparison reached with 40 eligible patients in the prospective part of the study can be assumed to be at least 80%.

Primary endpoint:

The primary endpoint (LPFS of MSCC) will be evaluated based on the sample size calculations. The evaluation will be performed in those patients, who are available for assessment of the primary endpoint and have received at least 80% of the planned RT dose. Due to the open nature of the study, a blind data review is not necessary. The safety population includes all patients who have received at least 1 fraction of high-precision RT.

LPFS is defined as freedom from progression of motor deficits during RT and freedom from an in-field recurrence of MSCC (i.e. freedom from motor deficits due to a recurrence of MSCC in the previously irradiated parts of the spine) following RT. Deterioration of motor deficits during RT will be counted as LPFS of 0 months. Freedom from an in-field recurrence following RT will be referenced from the last day of RT. LPFS rates will be calculated for each potential prognostic factor using the Kaplan-Meier method. Differences between the Kaplan-Meier curves will be calculated with the log-rank test (univariate analysis). Factors that achieve significance (p<0.05) or show a trend (p<0.06) on univariate analysis will be additionally included in a multivariate analysis (Cox proportional hazards model).

Secondary endpoints:

The comparison of the high-precision RT group and the conventional RT group with respect to their effect on motor function and sensory function (improvement, no further progression, deterioration) will be evaluated with the ordered logit model adjusted for propensity score, because the data for the impact of RT on motor and sensory function are ordinal (-1 = deterioration, 0 = no further progression, 1 = improvement). An improvement or deterioration of the motor function will be defined as a change of at least 1 point on a 5-point scale. Post-RT ambulatory and sphincter dysfunction rates will be compared between both groups with the Chi-square test stratified for propensity score. Effect of RT on motor function, post-RT ambulatory rates, sensory function and sphincter dysfunction will be evaluated directly after RT and at 1, 3 and 6 months following RT in those patients who are alive and available for assessment. P-values of <0.05 are considered significant.

Overall survival (OS) will be counted from the last day of RT. OS rates will be calculated with the Kaplan-Meier-method. Differences between Kaplan-Meier curves will be analyzed with the log-rank test. Again, p-values of <0.05 are considered significant. Factors that achieve significance or show a trend (p<0.06) on univariate analysis will be included in a multivariate analysis (Cox proportional hazards model). The analysis of OS will be conducted in the intent-to-treat population.

Data regarding pain, quality of life and toxicity will only be assessed in the study group.

ELIGIBILITY:
Inclusion Criteria:

* Motor deficits of the lower extremities resulting from MSCC, which have persisted for no longer than 30 days
* Confirmation of diagnosis by magnetic resonance (MR) imaging (computed tomography (CT) allowed)
* Age 18 years or older
* Written informed consent
* Capacity of the patient to contract

Exclusion Criteria:

* Previous RT or surgery of the spinal areas affected MSCC
* Symptomatic brain tumor or symptomatic brain metastases
* Metastases of the cervical spine only
* Other severe neurological disorders
* Pregnancy, lactation period
* Indication for decompressive surgery of affected spinal areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Rades, Professor, Principal Investigator — Radiation Oncology, University of Lübeck, Lübeck, Germany
Locations (1):
- Department of Radiation Oncology, University of Lübeck and University Medical Center Schleswig-Holstein, Ratzeburger Allee 160, 23562 Lübeck, Germany, Lübeck, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rades D, Cacicedo J, Conde-Moreno AJ, Segedin B, Lomidze D, Ciervide R, Hollaender NH, Schild SE. Comparison of 5 x 5 Gy and 10 x 3 Gy for metastatic spinal cord compression using data from three prospective trials. Radiat Oncol. 2021 Jan 7;16(1):7. doi: 10.1186/s13014-020-01737-7. PMID 33413492
- [Derived] Rades D, Cacicedo J, Conde-Moreno AJ, Segedin B, But-Hadzic J, Groselj B, Kevlishvili G, Lomidze D, Ciervide-Jurio R, Rubio C, Perez-Romasanta LA, Alvarez-Gracia A, Olbrich D, Doemer C, Schild SE, Hollaender NH. Precision Radiation Therapy for Metastatic Spinal Cord Compression: Final Results of the PRE-MODE Trial. Int J Radiat Oncol Biol Phys. 2020 Mar 15;106(4):780-789. doi: 10.1016/j.ijrobp.2019.11.401. Epub 2019 Dec 5. PMID 31812719
- [Derived] Rades D, Cacicedo J, Conde-Moreno AJ, Doemer C, Dunst J, Lomidze D, Segedin B, Olbrich D, Hollander NH. High-precision radiotherapy of motor deficits due to metastatic spinal cord compression (PRE-MODE): a multicenter phase 2 study. BMC Cancer. 2017 Dec 4;17(1):818. doi: 10.1186/s12885-017-3844-x. PMID 29202720

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-precision RT 5x5 Gy in 1 Week
Started | 44
Completed | 40
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | High-precision RT 5x5 Gy in 1 Week
Number analyzed (Participants) | 44
Age, Customized [Count of Participants; unit: Participants]
  Age: <=65 years | 30
  Age: >=66 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  caucasian | 44
  other | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 20
  Spain | 12
  Slovenia | 9
  Georgia | 3
primary tumor type [Count of Participants; unit: Participants]
  breast cancer | 9
  prostate cancer | 3
  myeloma/lymphoma | 5
  lung cancer | 13
  other tumors | 14
interval from tumor diagnosis to MSCC [Count of Participants; unit: Participants]
  <=15 months | 23
  >15 months | 21
number of involved vertebrae [Count of Participants; unit: Participants]
  1-2 | 30
  >=3 | 14
other bone metastases [Count of Participants; unit: Participants]
  no | 10
  yes | 34
visceral metastases [Count of Participants; unit: Participants]
  no | 16
  yes | 28
time developing motor deficits [Count of Participants; unit: Participants]
  1-7 days | 14
  8-14 days | 10
  >14 days | 20
ambulatory status [Count of Participants; unit: Participants]
  not ambulatory | 18
  ambulatory | 26
Eastern Cooperative Oncology Group performance score [Count of Participants; unit: Participants] — Performance status was rated with the Eastern Cooperative Oncology Group (ECOG), ranging from 0 to 5 (lower grade=better performance status).
  0: Fully active without restrictions.
  1. Restricted in physically strenuous activity; ambulatory and able to perform light or sedentary work.
  2. Ambulatory and capable of all self-care; unable to work; up and about >50% of hours awake.
  3. Capable of limited self-care; confined to bed/chair >50% of hours awake.
  4. Completely disabled. Totally confined to bed or chair.
  5. Dead.
  [Oken et al., Am J Clin Oncol 1982;5:649-55.]
  Participants
    ECOG 1-2 | 20
    ECOG 3-4 | 24
motor function [Count of Participants; unit: Participants]
  ambulatory without aid | 15
  ambulatory with aid | 12
  not ambulatory | 15
  complete paraplegia | 2
sensory function [Count of Participants; unit: Participants]
  absent | 0
  impaired | 17
  normal | 23
  unclear | 4
sphincter dysfunction [Count of Participants; unit: Participants]
  no | 37
  yes | 6
  unclear | 1
Distress (measured with the distress-thermometer) [Count of Participants; unit: Participants] — Distress (as an indicator of impairment of quality of life) was measured with the distress-thermometer. The patients rated their level of distress on a scale ranging from 0 (no distress) to 10 (extreme distress). Patients rated the distress they experienced during the last week and stated the reasons for distress from a list of items.
  [Holland JC, et al. J Natl Comp Cancer Network 2013;11:190-209.]
  Participants
    0-1 points | 1
    2-4 points | 11
    5-7 points | 15
    8-10 points | 16
    not available | 1
Pain (measured with a numeric self-rating scale) [Count of Participants; unit: Participants] — Pain was measured with a numeric self-rating scale ranging from 0 (no pain) to 10 (worst pain).
  Participants
    0-1 points | 8
    2-4 points | 11
    5-7 points | 14
    8-10 points | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Alive at 6 Months After Radiotherapy Without Deterioration of Motor Function During (or Directly After) Radiotherapy and Freedom From In-field Recurrence of Metastatic Spinal Cord Compression Following Radiotherapy
Description: Local Progression Free Survival (LPFS) was defined as freedom from progression of motor deficits during or one month following radiotherapy and freedom from in-field recurrence of metastatic spinal cord compression (MSCC) following radiotherapy.
  An in-field recurrence was defined as a recurrence of MSCC associated with motor deficits in the region of the spinal cord that had been previously irradiated for MSCC.
  In case of clinical suspicion of sich a recurrence, a spinal MRI was performed to confirm the diagnosis. Time to in-field recurrence was calculated from the last day of radiotherapy, and the patients were followed for a maximum of 6 months after the end of radiotherapy. The values of 6-month LPFS were estimated using the Kaplan-Meier method.
Time Frame: 6 months after the end of radiotherapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- High-precision Radiotherapy 5x5 Gy in 1 Week: Patients with motor deficits of the lower extremities due to metastatic spinal cord compression (MSCC) will receive 5x5 Gy of high-precision RT in 1 week.
  High-precision radiotherapy 5x5 Gy in 1 week: Patients included in this study will receive a high-precision radiotherapy with 5x5 Gy in 1 week
Arm/Group | High-precision Radiotherapy 5x5 Gy in 1 Week
Number analyzed (Participants) | 40
percentage of participants | 95.0 [81.5 to 98.7]
Statistical Analysis 1: Comparison: High-precision Radiotherapy 5x5 Gy in 1 Week; historical control group treated with 5 x 4 Gy; Test type: Superiority — It was assumed that radiotherapy with 5x4 Gy results in 6-month LPFS of 67% and an increase by 20% is clinically relevant when using 5x5 Gy. For comparison of 5x5 Gy and a historical control (5x4 Gy), it was assumed that it can be performed with a simple Pearson-Chi-Square test (2-sided significance level of 5%, power of 79%) if 40 patients treated with 5x5 Gy and 400 patients of the control group qualified for Propensity-Score adjusted comparison, assuming 6-month LPFS rates of 87% and 67%; p < 0.05, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20; In a prospective study, 6-month LPFS rates were 86% after longer-course (mainly 3Gyx10) and 67% after short-course radiotherapy (mainly 4Gyx5) [Rades D, et al., Int J Radiat Oncol Biol Phys 2009;73:228-34.]. For sample size calculations, it was assumed that conventional radiotherapy with 4Gyx5 results in 6-month LPFS of 67% and that an increase by 20% is clinically relevant and realistic with 5Gyx5. A sample size of 40 eligible patients was required for the phase 2 trial assuming that that 6-month LPFS would be 87% and estimated with a precision of +/-20% expressed as the half length of the associated two-sided confidence interval (95%), and power of >=80%. For comparison of phase 2 cohort and historical control group, it was assumed that this could be performed with a simple Pearson-Chi-Square test using a two-sided significance level of 5% (10%) and a power of 79% (86%) if 40 patients received 5Gyx5 and N=400 of the control group qualified for Propensity-Score adjusted comparison

2. Secondary Outcome: Number of Participants Showing Improvement of Motor Deficits Following Radiotherapy (Best Response)
Description: Motor function was evaluated using the following scale. Improvement of motor function was defined as a decrease of at least 1 point.
  0 = Normal strength
  1. = Ambulatory without aid
  2. = Ambulatory with aid
  3. = Not ambulatory
  4. = Complete paraplegia
  [Tomita T, et al., Acta Radiol Oncol 1983;22:135-143.]
Time Frame: up to 6 months following radiotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | High-precision RT 5x5 Gy in 1 Week
Number analyzed (Participants) | 40
Participants
  improvement of motor function | 24
  no improvement of motor deficits | 16

3. Secondary Outcome: Number of Participants Showing Improvement of Sensory Function Following Radiotherapy (Best Response)
Description: Sensory function was evaluated with the following scale, modified in accordance to the classification of the American Spinal Injury Association.
  0 = Absent
  1. = Impaired
  2. = Normal
  9 = Cannot be assessed
  [Baskin DS. Spinal cord injury. In Evans RW (Ed.), Neurology and trauma, WB Saunders, Philadelphia;1996, pp. 276-299.]
Time Frame: up to 6 months following radiotherapy
Population: Patients who had sensory deficits prior to the start of radiotherapy.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Sensory Deficits at Baseline: Patients who had sensory deficits prior to the start of radiotherapy.
Arm/Group | Patients With Sensory Deficits at Baseline
Number analyzed (Participants) | 16
Participants
  improvement of sensory deficits | 8
  no improvement of sensory deficits | 8

4. Secondary Outcome: Number of Participants Showing Improvement of Sphincter Dysfunction Following Radiotherapy (Best Response)
Description: Sphincter dysfunction was rates as yes (presence of sphincter dysfunction) or no (absence of sphincter dysfunction).
Time Frame: up to 6 months following radiotherapy
Population: Patients who had a sphincter dysfunction prior to the start of radiotherapy.
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Sphincter Dysfunction at Baseline: Patients who had a sphincter dysfunction prior to the start of radiotherapy.
Arm/Group | Patients With Sphincter Dysfunction at Baseline
Number analyzed (Participants) | 6
Participants
  improvement | 2
  no improvement | 2
  post-treatment assessment not available | 2

5. Secondary Outcome: Number of Participants Who Were Alive at 3 Months Following Radiotherapy Without Deterioration of Motor Function During (or Directly Following) Radiotherapy and Freedom From In-field Recurrence of Metastatic Spinal Cord Compression Following Radiotherapy
Description: Local Progression Free Survival (LPFS) was defined as freedom from progression of motor deficits during or one month following radiotherapy and freedom from in-field recurrence of metastatic spinal cord compression (MSCC) following radiotherapy.
  An in-field recurrence was defined as a recurrence of MSCC associated with motor deficits in the region of the spinal cord that had been previously irradiated for MSCC.
  In case of clinical suspicion of sich a recurrence, a spinal MRI was performed to confirm the diagnosis. Time to in-field recurrence was calculated from the last day of radiotherapy. The values of 3-month LPFS were estimated using the Kaplan-Meier method.
Time Frame: 3 months after the end of radiotherapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-precision RT 5x5 Gy in 1 Week
Number analyzed (Participants) | 40
percentage of participants | 95 [82 to 99]

6. Secondary Outcome: Number of Participants Who Were Alive at 6 Months Following Radiotherapy
Description: Overall Survival (OS) was defined as freedom from death of any cause. Time to death was calculated from the last day of radiotherapy, and the patients were followed for a maximum of 6 months after the end of radiotherapy. The values of 6-month OS were estimated using the Kaplan-Meier method.
Time Frame: 6 months after the end of radiotherapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-precision RT 5x5 Gy in 1 Week
Number analyzed (Participants) | 40
percentage of participants | 45.0 [26.7 to 57.6]

7. Secondary Outcome: Number of Participants Who Experienced Relief of Pain at 1 Month Following Radiotherapy Compared to Baseline
Description: Vertebral pain was measured with a numeric self-rating scale ranging from 0 (no pain) to 10 (worst pain).
  Pain relief was defined as improvement (=decrease of pain) by at least 2 points without increase of analgesics. Patients with baseline-scores of 0-1 points were not included, since improvement by 2 points was not possible.
Time Frame: Evaluation at 1 month following radiotherapy
Measure: Count of Participants; unit: Participants
Groups:
- Patients With a Pain Score of >1 at Baseline: Patients who had a pain score of >1 prior to the start of RT and were evaluable for pain relief at 1 month following RT.
Arm/Group | Patients With a Pain Score of >1 at Baseline
Number analyzed (Participants) | 21
Participants
  pain relief | 13
  no pain relief | 8

8. Secondary Outcome: Number of Participants Who Experienced Relief of Distress at 1 Month Following Radiotherapy Compared to Baseline
Description: Distress (as an indicator of impairment of quality of life) was measured with the distress-thermometer. the patients rated their level of distress on a scale ranging from 0 (no distress) to 10 (extreme distress). Patients rated the distress they experienced during the last week and stated the reasons for distress from a list of items.
  An improvement (lower score) by 2 points was considered a clinically relevant relief of distress. Patients with baseline-scores of 0-1 points were not included, since improvement by 2 points was not possible.
Time Frame: Evaluation at 1 month following radiotherapy
Measure: Count of Participants; unit: Participants
Groups:
- Patients With a Distress Score of >1 at Baseline: Patients who had a distress score of >1 prior to the start of RT and were evaluable for relief of distress at 1 month following RT.
Arm/Group | Patients With a Distress Score of >1 at Baseline
Number analyzed (Participants) | 24
Participants
  relief of distress | 13
  no relief of distress | 11

9. Secondary Outcome: Number of Participants Experiencing at Least One Grade >=2 Radiotherapy-related Toxicity
Description: Toxicity was assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) (version 4)
Time Frame: during radiotherapy and up to 6 months following radiotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | High-precision RT 5x5 Gy in 1 Week
Number analyzed (Participants) | 40
Participants
  grade 2-3 toxicity: toxicity | 4
  grade 2-3 toxicity: no toxicity | 36
  grade 3 toxicity: toxicity | 1
  grade 3 toxicity: no toxicity | 39

10. Secondary Outcome: Number of Participants Who Were Able to Walk Following Radiotherapy
Description: Ambulatory status was assessed using the following scoring system:
  0=Normal strength
  1. Ambulatory without aid
  2. Ambulatory with aid
  3. Not ambulatory
  A patient with a score equal to or less than 2 is considered "able to walk". Both participants that could and could not walk prior to radiotherapy have been included in this assessment.
Time Frame: up to 6 months following radiotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | High-precision RT 5x5 Gy in 1 Week
Number analyzed (Participants) | 40
Participants
  able to walk following radiotherapy | 33
  not able to walk following radiotherapy | 7

ADVERSE EVENTS:
Time Frame: during the period of radiotherapy and up to 6 months during the period of follow up
Arm/Group | High-precision RT 5x5 Gy in 1 Week
All-Cause Mortality (participants affected / at risk) | 22/40
Serious Adverse Events (participants affected / at risk) | 5/40
Other Adverse Events (participants affected / at risk) | 10/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-precision RT 5x5 Gy in 1 Week (N=40)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Heart failiure (Cardiac disorders) | 1 (1)
Unknown death (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Systemic aspergillosis (Infections and infestations) | 1 (1)
Pulmonary embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-precision RT 5x5 Gy in 1 Week (N=40)
Nausea (Gastrointestinal disorders) | 10 (17)
Diarrhea (Gastrointestinal disorders) | 7 (13)
Fatigue (General disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT03070431/Prot_SAP_ICF_000.pdf